CLINICAL TRIAL: NCT04242524
Title: The Impact of Bariatric Surgery on Adipocyte Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB14-0984
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: insulin; adipocyte; gene expression
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Circadian Clock Alignment - High BMI (Experimental): Subjects will come to the Sleep Lab three nights before their bariatric surgery procedure for an intervention that will align their central circadian clock. The intervention includes eating meals and snacks at fixed times and having lights off at a specific time at night and lights on at a specific time in the morning.
  Interventions: Behavioral: Circadian Clock Alignment
- Circadian Clock Control - High BMI (Active Comparator): Subjects will not come to the Sleep Lab and will live normally at home with no changes to their meal, sleep or wake times.
  Interventions: Behavioral: Circadian Clock Control
- Circadian Clock Control - Low BMI (Active Comparator): Subjects will not come to the Sleep Lab and will live normally at home with no changes to their meal, sleep or wake times.
  Interventions: Behavioral: Circadian Clock Control

INTERVENTIONS:
Behavioral: Circadian Clock Alignment — Use timed lights and meals to align the circadian clock
  Arms: Circadian Clock Alignment - High BMI
Behavioral: Circadian Clock Control — No circadian clock alignment
  Arms: Circadian Clock Control - High BMI; Circadian Clock Control - Low BMI

SUMMARY:
The purpose of this study is to understand how daily rhythms of behavior affect the expression of genes in fat cells, and how these daily cycles affect the way fat cells respond to insulin (a hormone that controls blood sugar levels) before and after bariatric surgery.

DETAILED DESCRIPTION:
Bariatric surgery as a means of weight loss has become increasingly popular over the last 10-15 years. In addition to promoting weight loss, bariatric surgery has become increasingly recognized for use in the management of diabetes. Recent studies have indicated that bariatric surgery can result in a marked improvement in insulin sensitivity before long term weight loss is attained. The goal of this project is to delineate the changes in the insulin responsiveness of subcutaneous adipocytes obtained by needle biopsy 2 weeks prior to surgery vs. 12 weeks after bariatric surgery, which could account for improvements in overall insulin sensitivity seen before any long-term sustained weight loss has occurred. The investigators will also examine gene expression in adipocytes (fat cells).

ELIGIBILITY:
Obese Subjects

Inclusion Criteria:

* 18-55 years old
* Female
* BMI greater than 40 kg/m2
* Scheduled for bariatric surgery at the Center for the Surgical Treatment of Obesity at the University of Chicago
* Signed informed consent

Exclusion Criteria:

* Male
* Diagnosed with a systemic illnesses, including heart, renal, liver, or malignant disease
* Uncontrolled hypertension (blood pressure greater than 140 mmHg systolic and 90 mmHg diastolic without medication)
* use of beta blockers
* hemoglobin less than 11.5g/dL
* known allergy to lidocaine
* pregnancy
* lactation
* Subjects will not have undergone surgery, donated a unit of blood, or participated in another clinical study within the last 4 weeks prior to consent.
* Post-menopausal

Non-Obese Subjects

Inclusion Criteria:

* 18-55 years old
* Female
* BMI less than 30 kg/m2
* Signed informed consent

Exclusion Criteria:

* Male
* Diagnosed with a systemic illnesses, including heart, renal, liver, or malignant disease
* Uncontrolled hypertension (blood pressure greater than 140 mmHg systolic and 90 mmHg diastolic without medication)
* use of beta blockers
* hemoglobin less than 11.5g/dL
* known allergy to lidocaine
* pregnancy
* lactation
* Subjects will not have undergone surgery, donated a unit of blood, or participated in another clinical study within the last 4 weeks prior to consent.
* Post-menopausal

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 82 (Estimated)
Dates: Start 2015-03-26 (Actual); Primary Completion 2025-12 (Actual); Study Completion 2025-12 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | 12 weeks
  Insulin sensitivity will be measured as the by the phosphorylation level of Akt in adipocytes (fat cells) at baseline and 12 weeks post bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brady, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no IRB approval or plan to make IPD available to other researchers.